CLINICAL TRIAL: NCT02491320
Title: Effect of Acupuncture Pre-treatment Combined With Letrozole on Live Birth in Infertile Women With Polycystic Ovary Syndrome
Brief Title: The Clinical Trial of Acupuncture Pre-treatment on PCOS
Acronym: PCOSAPct
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: The University of Hong Kong (Other); Karolinska Institutet (Other); Xuzhou Maternity and Child Health Care Hospital (Other); Hexian Memorial Affiliated Hospital of Southern Medical University (Unknown)
Responsible Party: Principal Investigator, Hongxia Ma, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOSAPct
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; acupuncture; pre-treatment; Letrozole; Live Birth
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Treatment Expectations; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-treatment acupuncture + letrozole (Experimental): A 16 week acupuncture pretreatment followed by letrozole(LE). Acupuncture treatment will start on day 3-5 after a spontaneous period or after a withdrawal bleeding following progestin. All subjects will be requested to use contraception during the 16 week acupuncture pretreatment. They will receive acupuncture treatment three times a week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 16 weeks. After 16 weeks of acupuncture treatment, LE will start on day 2-3 after a spontaneous period or after a withdrawal bleeding after progestin administration. The subjects will be instructed to have intercourse on a regular basis during the cycles.
  Interventions: Other: Pre-treatment acupuncture; Drug: Letrozole
- Letrozole (Active Comparator): LE alone. LE will be started on day 3-5 after a spontaneous period or a withdrawal bleeding following progestin. The subjects will be instructed to have intercourse on a regular basis during the cycles.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Other: Pre-treatment acupuncture — Acupuncture treatment will start on day 3-5 after a spontaneous period or after a withdrawal bleeding following progestin. They will receive acupuncture treatment three times a week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 16 weeks.
  Other Names: Pretreatment
  Arms: Pre-treatment acupuncture + letrozole
Drug: Letrozole — Starting from 2.5mg daily from day 3-5 for 5 days after a spontaneous period or after a withdrawal bleeding following progestin, one time per day.Participants are treated for up to 4 cycles.
  Other Names: Letrozole(Femara, Novartis Pharmaceuticals)

SUMMARY:
This is a study protocol for a multicenter, randomized, and controlled trial. In this protocol, we present a randomized controlled trial comparing acupuncture pretreatment followed by letrozole vs letrozole alone in polycystic ovary syndrome (PCOS) women with anovulatory infertility. The high prevalence of insulin resistance (IR) in women with PCOS women is considered to be one of the major pathophysiological changes of PCOS, leading to anovulatiory infertility. A study has shown that electro-acupuncture could significantly improve insulin sensitivity. The effect of acupuncture pretreatment on anovulatory PCOS women followed by ovulation induction has not been investigated before. A total of 384 patients enrolled in this study will be randomized into one of two groups. The treatment group: a 16 week acupuncture pretreatment followed by 4 cycles of letrozole and the control group: 4 cycles of letrozole alone. The primary outcome is the live birth rate. We postulate that acupuncture pretreatment followed by letrozole results in a higher live birth rate when compared with letrozole alone.

DETAILED DESCRIPTION:
1. Study content 1.1 Study design This is a multi-centered, randomized, clinical trial. 1.2 Subject selection and exclusion

Initially, 384 PCOS women anovulatory infertility will be recruited from four hospitals in mainland China: Department of Traditional Chinese Medicine in the first affiliated hospital of Guangzhou Medical University, Department of Gynecology in Xuzhou maternity & child health hospital, Department of Reproduction in Dalian Municipal Women and Children's Medical Center, and Department of Traditional Chinese Medicine in Hexian memorial affiliated hospital of Southern Medical University if they meet the inclusion criteria and do not have the exclusion criteria. Eligible subjects will be approached and sign the consent form after detailed explanation and counseling. Recruited subjects will be randomized to one of two groups:

Treatment group: a 16 week acupuncture pre-treatment followed by LE and Control group: LE alone 1.3 Screening visit 1.3.1 Obtain signed informed consent 1.3.2 Complete physical examination Perform complete physical examination including height, weight, hip and waist measurement. Height and weight will be recorded to the nearest 0.1 cm and 0.1 kg respectively. Waist and hip circumference will be recorded to the nearest 1 cm. And assessment of hirsutism by Ferriamn Gallwey score (FG), acne standard acne lesion counts, and pelvic exam with Pap smear or TCT.

1.3.3 Perform transvaginal ultrasound of the uterus and ovaries

1. Uterus, including the uterine dimensions, endometrial thickness and echo type, other uterine abnormalities, presence and size of leiomyoma will be obtained through transvaginal ultrasound.
2. Ovaries, including the ovarian size in three dimensions, the size of the largest ovarian follicle/cyst and size of every follicle with a mean diameter greater than 10 mm, and total antral follicle (small follicles with mean diameter < 10 mm) count of each ovary will be obtained through transvaginal ultrasound.

1.3.4 Check urine pregnancy test 1.3.5 Laboratory Examination

1. Serum levels of sex hormone steroids including blood follicle-stimulating hormone (FSH), luteinizing hormone (LH), estrogen (E2), prolactin (PRL) and T, free testosterone, sex hormone binding globulin (SHBG), and thyroid stimulating hormone (TSH) will be evaluated on the second day of the spontaneous period or a withdrawal bleeding.
2. Fasting blood was taken to determine the examination of metabolic and safety profile, including fasting blood glucose, insulin, C-peptide, HbA1c, triglycerides, total cholesterol, high density lipoprotein (HDL-C), low density lipoprotein (LDL-C), CBC, Renal, and Liver Profile.
3. The oral glucose tolerance test (OGTT) with 75 g glucose will be performed in all subjects after an overnight fast. Blood samples will be obtained to measure plasma glucose and serum insulin at 0, 60, and 120 min during the OGTT.

1.3.6 Complete questionnaires Quality of life will be assessed by the short form 36(SF-36), the Chinese Quality of Life (ChiQOL), sleeping questionnaires and the Polycystic Ovary Syndrome Questionnaire (PCOS-QOL). Investigators will also assess symptoms of anxiety and depression by the Zung SAS and Zung SDS questionnaires. And complete the quantization table of traditional Chinese medicine (TCM) syndromes about PCOS.

1.3.7 Exclusion of other infertility factors of the couple The semen analysis of the husband and tubal patency of the patient will be assessed.

1.3.8 Preconception counseling Complete the questionnaire of risk factors for genetic disorders, TORCH screening (Toxoplasmosis, Rubella, Cytomegalo Virus, and Herpes Virus) and HIV screening, and folic acid prescription.

1.3.9 Progestin withdrawal Provide progestin prescription to induce withdrawal bleed, with instructions to begin medication once eligibility is determined.

1.4 Baseline visit 1.4.1 Distribute home pregnancy test 1.4.2 Distribute folate 1.4.3 Distribute intercourse and menstrual journal logs 1.4.4 Take blood sample for repository and DNA Collect 20ml blood, and distributed store 10ml blood after serum separation. Other 10ml blood is for determination of DNA.

1.5 Intervention arms

Eligible patients will be randomized into one of the two arms:

Treatment group: i.e. a 16 week acupuncture pretreatment followed by LE. Acupuncture treatment will start on day 3-5 after a spontaneous period or after a withdrawal bleeding following progestin. All subjects will be requested to use contraception during the 16 week acupuncture pretreatment. They will receive acupuncture treatment three times a week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 16 weeks. After 16 weeks of acupuncture treatment, LE will start on day 2-3 after a spontaneous period or after a withdrawal bleeding after progestin administration. The subjects will be instructed to have intercourse on a regular basis during the cycles.

Control group: i.e. LE alone. LE will be started on day 3-5 after a spontaneous period or a withdrawal bleeding following progestin. The subjects will be instructed to have intercourse on a regular basis during the cycles.

1.5.1 Acupuncture protocol Investigators base the rationale of acupuncture protocols on Western Medical theories and the study protocol follows the CONSORT and STRICTA recommendations with detailed descriptions of the treatment including number of needle used, how needles will be stimulated (manual, electrical), frequency of sessions, and length of treatment period. Investigators will use fixed acupuncture protocols.

Disposable, single-use, sterilized needles made of stainless steel, 0.25 x 30 mm and 0.30 x 40/50 mm (Hwoto, Suzhou Medical Appliance Fact. 215005 Suzhou, China) will be inserted to a depth of 15-35 mm in segmental acupuncture points located in abdominal and leg muscles with innervations corresponding to the ovaries. Two sets of acupuncture points will be alternated every second treatment. The first set consists of conception vessel (CV) 3, CV 12, and stomach (ST) 29 bilaterally and in the muscles above the knee, ST 34, and ST 33 bilaterally and below the knee, spleen (SP) 6 and ST 36. Needles will also be placed in extra segmental acupuncture points that do not innervate the ovaries large intestine (LI) 4 bilaterally. In total 14 needles will be placed and all will be stimulated manually by rotating the needle to evoke needle sensation (de qi) once when inserted. The following points will be connected to an electrical stimulator (Export Abteilung, Schwa-Medico GmbH, Wetzlarer Str. 41-43; 35630 Ehringshausen): CV 3 to CV 12, ST 29 bilateral, and ST34 to ST 33 bilateral. Stimulation are given as low-frequency EA of 2Hz, 0.3 ms pulse length and with an intensity adjusted to produce local muscle contractions without pain or discomfort. Needles not connected to the electrical stimulator will be manually stimulated to evoke needle sensation every 10 min, in total 4 times. The second set consists of 14 needles placed in segmental abdominal points and stimulated electrically: ST 27 bilaterally, CV6 connected to CV10; and leg points: SP10 connected to a non-acupuncture point located 6 cun proximal of patellas medial border (electrical stimulation), and SP 6 and liver (LR) 3 bilaterally (manual stimulation). Extra segmental points are pericardium (PC) 6 bilaterally (manual stimulation).

1.5.2 Needle insertion technique Needle insertion should be gentle. Tighten the skin by pressing around the area of needle insertion and gently insert the needle. Don't do it too quickly, be gentle.

1.5.3 Needles and stimulation Needles are for single use. Needle size: 0.25x30 mm or 0.30 x 40 or 0.30 x 50 mm. Select needle length with respect to the patients BMI. If the patient has a low BMI and is thin use the 0.25 x 30 mm needle. If the patient is overweight, use the 0.30 x 40 mm needles. Obese patients, use needle with the size 0.30 x 50 or 75 mm. Depth of insertion may vary from patient to patient. They should be placed with a depth deep enough to reach muscle/fibrous tissue. When needle are inserted, stimulate the needle gently until de qi (needle sensation reflecting activation of sensory afferents). As soon as de qi has been reached, make sure that the needle doesn't hurt or cause any pain and discomfort.

Attach the electrodes according to the protocol. Turn on the stimulator (program 10) and increase the intensity. Instructions to the patient: "As high as possible but with no pain or discomfort". Don't start with too intensive stimulation. After 10 minutes, stimulate needles without electricity and ask if the intensity of the electrical stimulation is ok, or if it should be increased/decreased. Repeat after 20 minutes and again after 30 minutes. Turn off the stimulator and release the patient.

1.5.4 Acupuncture treatment

1. Record time of the day and acupuncturist name when the patient receives acupuncture.
2. Note the intensity of stimulation (mA). It may vary between the different electrodes. Note the range e.g. 1.2 - 3.0 mA.
3. Note any other events that may affect the treatment (positive or negative).
4. Note concomitant medications.
5. Collect menstrual and intercourse journal logs at the end of every cycle.
6. Check urine pregnancy test before each acupuncture treatment. If pregnancy test is positive, no acupuncture treatment should be performed.

1.5.5 Letrozole After 16 weeks of acupuncture pretreatment, which the patients in the intervention group and the patients in the control group will receive LE (Femara, Novartis Pharmaceuticals), starting from 2.5mg daily from day 2-3 for 5 days after a withdrawal bleeding. Participants are treated for up to 4 cycles. If the patient is pregnant, the treatment should be stopped.

If there is evidence of ovulation (i.e. serum progesterone level on the 3th week was higher than 3 ng/mL) or delayed one week, this dose will be maintained. In patients with no ovulatory response, the dose will be increased to LE 5mg a day for five days until LE 7.5 mg per day for five days will be reached. The same LE dose will be continued in the next cycle if the patients are shown to be ovulating. And the maximum daily dose of LE is 7.5 mg (three pills) daily.

1.6 Monitoring and examination during the treatment And all subjects will be instructed to have intercourse on a regular basis during the entire study period. The optimal frequency will be once every 2-3 days. Urine pregnancy test will be checked before each acupuncture treatment of ovulation. And serum progesterone level test will be checked in the local lab at day on the 3th week of the first cycle and every week of the last three cycles.

The transvaginal ultrasound exam will take place in the anticipated luteal phase of the cycle, and initially will be scheduled 3 weeks after the initiation of medication, with a window of 4 days on either side of this day (i.e. Day 17-25, assuming a Day 3 medication start, or Day 19-27, assuming a Day 5 start). The ultrasound includes the endometrial thickness and echogenicity, as well as the number, size, and echogenic characteristics of follicles/cysts on the ovary (including an antral follicle count).

Investigators can decide whether the patients have the ovulation respond based on the results of serum progesterone level and transvaginal ultrasound. There will be three possible scenarios: ovulation, ovulation delay and non-ovulation. 1) Ovulation, i.e. serum progesterone level on the 3th week was higher than 3 ng/mL, and ultrasound may provide presumptive evidence of ovulation. Check urine pregnancy test to exclude pregnancy and start with LE tablet on day 3-5 of menstruation, and the dose of which will be maintained; 2) Ovulation delay, P<3 ng/mL, but the ultrasound will show there is evidence of follicular development, (i.e. a follicle with a mean diameter ≥12 mm). Investigators can wait for one more week and continue the acupuncture treatment. Check urine pregnancy test to exclude pregnancy and start with LE tablet on day 3-5 of menstruation, and the dose of which will be maintained; 3) Non-ovulation, P<3 ng/mL, and the ultrasound will not found any follicle with a mean diameter ≥12 mm. The patient will also receive LE tablet on day 3-5 of her cycle, and she will be instructed to increase her study drug by one tablet per day for five days.

Every menstruation should be detailed recorded, including the date, volume and duration of menstruation.

1.7 End of pre-treatment visit

1) Repeat OGTT. 2) Collect menstrual journal logs. 1.8 Pregnancy visit(only with conception)

1. Complete adverse event query.
2. Take blood for serum quantitative hCG levels until the ultrasound can observe the gestational sacs (1500-2000IU/ml).
3. Perform transvaginal ultrasound for the number of gestational sacs, location, dimensions, presence and size of fetal parts, and documentation of visualization of fetal heart motion, documentation of any pregnancy related abnormalities when hCG levels or clinical manifestations appear as pregnancy.

1.9 End of treatment visit

1. Perform physical examination, including vital signs, height, weight, hip and waist measurements as well as repeating hirsutism and acne assessments after the end of treatment or pregnancy.
2. Repeat the serum levels of sex hormone steroids and metabolic profile.
3. Repeat OGTT.
4. Collect 20ml blood, and distributed store 10ml blood after serum separation. Other 10ml blood is for determination of DNA.
5. Repeat QOL, sleeping, anxiety/depression questionnaires, and the quantization table of TCM.
6. Collect menstrual and intercourse journal logs.
7. Record adverse events and concomitant medications.
8. Arrange follow up for subjects who have conceived and obtain release of records for pregnancy and neonatal records.

1.10 Follow up visit For those women who have an ongoing pregnancy, arrangements will be made to follow the outcome of the pregnancy at the end of first trimester and also after delivery or termination of gestation. All pregnancies (including multiples) will be followed to monitor the weight, glucose tolerance, blood pressure and fetal growth and to determine the abortion rate, complication rates and pregnancy outcomes. The glucose tolerance will be test by glucose screening test with 75 g glucose performed in all pregnancies at 24-28 weeks of pregnancy. Patients will be informed to notify study personnel of the outcome of the pregnancy and investigators will obtain release of record forms from treating physicians to obtain copies of relevant medical records. Delivery records of both mother and newborn will be requested to determine the birth weight, length of gestation, and any prenatal complication of mother or neonatal complication of the infant. Phone contacts will be initiated if the patient has not contacted study personnel by six weeks beyond the original estimated date of confinement.

And investigators will collect pregnancy outcome data. Investigators will track the outcomes of all subjects who have a positive serum pregnancy screen during the course of this study. Investigators will record biochemical pregnancies (defined as positive serum pregnancy screens without ultrasonically detected pregnancies), ectopic pregnancies, and all intrauterine pregnancy losses both before and after 20 weeks including missed abortions, spontaneous abortions, elective abortions, fetal demises, and stillbirths. Investigators will review pregnancy and birth records of the mother and of the fetus to establish neonatal morbidity and mortality and the presence of fetal anomalies. Investigators will extract from these records concomitant medical and obstetrical conditions, exposure information on all other medical products used, including prescription products, over-the-counter (OTC) products, dietary supplements, vaccines, and insertable or implantable medical devices. Investigators will file individual case reports for all congenital anomalies, which will be considered a serious adverse event.

1.11 Safety analysis Adverse events will be categorized and percentage of patients experiencing adverse events and serious adverse events during the treatment period will be documented. Chi-square tests will be performed to examine differences in the proportion of total and categories of adverse events.

1.12 Statistical tests One sample of the Kolmogorov-Smirnov test will be used to test the normal distribution of continuous variables. Continuous variables will be shown as means ± standard deviations if they are normally distributed or as medians with interquartile ranges if they are not normally distributed. Statistical comparison will be carried out according to the intention to treat by Student's t-test, Mann-Whitney U-test, and Wilcoxon signed ranks test for continuous variables and by χ2 tests for categorical variables where appropriate. All statistical analyses of the data will be performed using the SPSS program version 21.0 (SPSS Inc., Chicago, IL, USA), and a P-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 20 and 40 years.
2. Confirmed diagnosis of PCOS according to 2003 modified Rotterdam criteria
3. According to World Health Organization standards (2010), semen analysis of the husband must meet ① or ②. ①sperm concentration ≥15*106/ml and total motility ≥40% . ② Total motile sperm count ≥9 million, i.e. semen volume*sperm density*percentage of motile sperm ≥9 million.
4. At least one patent tube shown by hysterosalpingogram or diagnostic laparoscopy. The results will be valid for 3 years if the patients do not have a history of abortion or pelvic operation.

Exclusion Criteria:

1) Exclusion of other endocrine disorders:

* Patients with hyperprolactinemia (defined as two prolactin levels at least one week apart 25 ng/mL or greater or as determined by local normative values). The goal of eliminating patients with documented hyperprolactinemia is to decrease the heterogeneity of the PCOS population. These patients may be candidates for ovulation induction with alternate regimens (dopamine agonists). A normal level within the last year or on treatment is adequate for entry.

  * Patients with FSH levels > 15 mIU/mL. A normal level within the last year is adequate for entry.

    * Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or >5.5 mIU/mL). A normal level within the last year is adequate for entry.

      * Patientsdiagnosed with Type I or Type II diabetes who are poorly controlled (defined as a Hb A1c level > 7.0%), or patients receiving antidiabetic medications such as insulin, thiazolidinediones, acarbose, or sulfonylureas likely to confound the effects of study medication; Patients currently receiving metformin XR (extended release) for a diagnosis of Type I or Type II diabetes or for PCOS are also specifically excluded.

        ⑤Patients with suspected Cushing's syndrome. 2) Use of hormonal or other medication including Chinese Herbal prescriptions which may affect the outcome at least in the past 2 months.

        3) Acupuncture the last 2 months. 4) Pregnancy within the past 6 weeks. 5) Within 6 weeks post-abortion or postpartum. 6) Breastfeeding within the last 6 months. 7) Not willing to give written consent to the study. 8) Additional exclusion criteria

        1. Patients with a suspected adrenal or ovarian tumor secreting androgens. 2. Couples with previous sterilization procedures (vasectomy, tubal ligation) which have been reversed. The prior procedure may affect study outcomes, and patients with both a reversed sterilization procedure and PCOS are rare enough that exclusion should not adversely affect recruitment.

        3. Subjects who have undergone a bariatric surgery procedure in the recent past (<12 months) and are in a period of acute weight loss or have been advised against pregnancy by their bariatric surgeon.

        4. Patients with untreated poorly controlled hypertension defined as a systolic blood pressure 160 mm Hg or a diastolic 100 mm Hg obtained on two measures obtained at least 60 minutes apart.

        5. Patients with known congenital adrenal hyperplasia. 6. Patients on oral contraceptives, depot progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive forms or implants, especially where the implants are still in place. A one-month washout will be required for patients on oral cyclic progestins.

        7. Patients with liver disease defined as AST or ALT > 2 times normal or totalbilirubin >2.5 mg/dL. Patients with renal disease defined as BUN > 30 mg/dL or serum creatinine> 1.4 mg/dL.

        8. Patients with significant anemia (Hemoglobin < 10 g/dL). 9. Patients with a history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident.

        10. Patients with known heart disease that is likely to be exacerbated by pregnancy.

        11. Patients with a history of, or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma. A normal Pap smear or TCT result will be required for women 21 and over.

        12. Patients with a current history of alcohol abuse. Alcohol abuse is defined as >14 drinks/week or binge drinking.

        13. Patients enrolled simultaneously into other investigative studies that require medications, proscribe the study medications, limit intercourse, or otherwise prevent compliance with the protocol.

        14. Patients who anticipate taking longer than a one month break during the protocol should not be enrolled.

        15. Patients taking other medications known to affect reproductive function or metabolism. These medications include oral contraceptives, GnRH agonists and antagonists, antiandrogens, gonadotropins, anti-obesity drugs, Chinese herbal formula, anti-diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, ACE inhibitors, and calcium channel blockers. The washout period on all these medications will be two months.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Up to 18 months
  Live birth rate

SECONDARY OUTCOMES:
Ovulation rate | Up to 8 months
  Ovulation rate
Ongoing pregnancy rate | Up to 11 months
  Ongoing pregnancy rate
Multiple pregnancy rates | Up to 18 months
  Multiple pregnancy rates
Miscarriage rate | Up to 11 months
  Loss of an intrauterine pregnancy before 20 completed weeks of gestation
Pregnancy complications rate | Up to 18 months
  Pregnancy complications rate
Hormonal profile | Up to 8 months
  FSH, LH, T, SHBG and DHEAS
Metabolic profile | Up to 8 months
  Glucose and insulin concentrations, C-peptide, HbA1c, cholesterol, triglycerides, HDL-C and LDL-C
HOMA-IR | Up to 8 months
  HOMA-IR
Body composition(a composite) | Up to 8 months
  Weight, BMI, waist-to-hip circumference, FG and acne lesion counts
Questionnaires(a composite) | Up to 8 months
  SF-36, ChiQOL, sleeping questionnaires, PCOS-QOL, Zung SAS, Zung SDS questionnaires and the quantization table of TCM syndromes about PCOS.
Side effect profile | Up to 18 months
  Side effect profile
AUCglu | Up to 8 months
  AUCglu
AUCins | Up to 8 months
  AUCins

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Ma, PhD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Juan Li, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Elisabet Stener-Victorin, PhD, Principal Investigator — Karolinska Institutet; Ernest HY NG, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ghazeeri G, Kutteh WH, Bryer-Ash M, Haas D, Ke RW. Effect of rosiglitazone on spontaneous and clomiphene citrate-induced ovulation in women with polycystic ovary syndrome. Fertil Steril. 2003 Mar;79(3):562-6. doi: 10.1016/s0015-0282(02)04843-4. PMID 12620440
- [Background] Katulski K, Czyzyk A, Podfigurna-Stopa A, Genazzani AR, Meczekalski B. Pregnancy complications in polycystic ovary syndrome patients. Gynecol Endocrinol. 2015 Feb;31(2):87-91. doi: 10.3109/09513590.2014.974535. Epub 2014 Oct 30. PMID 25356655
- [Background] Wolf LJ. Ovulation induction. Clin Obstet Gynecol. 2000 Dec;43(4):902-15. doi: 10.1097/00003081-200012000-00020. PMID 11100305
- [Background] Legro RS, Brzyski RG, Diamond MP, Coutifaris C, Schlaff WD, Casson P, Christman GM, Huang H, Yan Q, Alvero R, Haisenleder DJ, Barnhart KT, Bates GW, Usadi R, Lucidi S, Baker V, Trussell JC, Krawetz SA, Snyder P, Ohl D, Santoro N, Eisenberg E, Zhang H; NICHD Reproductive Medicine Network. Letrozole versus clomiphene for infertility in the polycystic ovary syndrome. N Engl J Med. 2014 Jul 10;371(2):119-29. doi: 10.1056/NEJMoa1313517. PMID 25006718
- [Background] DeUgarte CM, Bartolucci AA, Azziz R. Prevalence of insulin resistance in the polycystic ovary syndrome using the homeostasis model assessment. Fertil Steril. 2005 May;83(5):1454-60. doi: 10.1016/j.fertnstert.2004.11.070. PMID 15866584
- [Background] Legro RS, Castracane VD, Kauffman RP. Detecting insulin resistance in polycystic ovary syndrome: purposes and pitfalls. Obstet Gynecol Surv. 2004 Feb;59(2):141-54. doi: 10.1097/01.OGX.0000109523.25076.E2. PMID 14752302
- [Background] Homburg R. Clomiphene citrate--end of an era? A mini-review. Hum Reprod. 2005 Aug;20(8):2043-51. doi: 10.1093/humrep/dei042. Epub 2005 May 5. PMID 15878925
- [Background] Stener-Victorin E, Waldenstrom U, Tagnfors U, Lundeberg T, Lindstedt G, Janson PO. Effects of electro-acupuncture on anovulation in women with polycystic ovary syndrome. Acta Obstet Gynecol Scand. 2000 Mar;79(3):180-8. PMID 10716298
- [Background] Johansson J, Redman L, Veldhuis PP, Sazonova A, Labrie F, Holm G, Johannsson G, Stener-Victorin E. Acupuncture for ovulation induction in polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2013 May 1;304(9):E934-43. doi: 10.1152/ajpendo.00039.2013. Epub 2013 Mar 12. PMID 23482444
- [Background] Pastore LM, Williams CD, Jenkins J, Patrie JT. True and sham acupuncture produced similar frequency of ovulation and improved LH to FSH ratios in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Oct;96(10):3143-50. doi: 10.1210/jc.2011-1126. Epub 2011 Aug 3. PMID 21816787
- [Background] Lai MH, Ma HX, Yao H, Liu H, Song XH, Huang WY, Wu XK. [Effect of abdominal acupuncture therapy on the endocrine and metabolism in obesity-type polycystic ovarian syndrome patients]. Zhen Ci Yan Jiu. 2010 Aug;35(4):298-302. Chinese. PMID 21090334
- [Background] Jedel E, Labrie F, Oden A, Holm G, Nilsson L, Janson PO, Lind AK, Ohlsson C, Stener-Victorin E. Impact of electro-acupuncture and physical exercise on hyperandrogenism and oligo/amenorrhea in women with polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E37-45. doi: 10.1152/ajpendo.00495.2010. Epub 2010 Oct 13. PMID 20943753
- [Background] Zheng YH, Wang XH, Lai MH, Yao H, Liu H, Ma HX. Effectiveness of abdominal acupuncture for patients with obesity-type polycystic ovary syndrome: a randomized controlled trial. J Altern Complement Med. 2013 Sep;19(9):740-5. doi: 10.1089/acm.2012.0429. Epub 2013 May 15. PMID 23676106
- [Background] Xu J, Qu HQ, Fang HL. [Effect of electroacupuncture combined with auricular point tapping and pressing on serum insulin and testosterone in the patients of obese women with polycystic ovary syndrome]. Zhongguo Zhen Jiu. 2009 Jun;29(6):441-3. Chinese. PMID 19563188
- [Background] Stener-Victorin E, Wu X. Effects and mechanisms of acupuncture in the reproductive system. Auton Neurosci. 2010 Oct 28;157(1-2):46-51. doi: 10.1016/j.autneu.2010.03.006. Epub 2010 Mar 29. PMID 20350839
- [Background] Raja-Khan N, Stener-Victorin E, Wu X, Legro RS. The physiological basis of complementary and alternative medicines for polycystic ovary syndrome. Am J Physiol Endocrinol Metab. 2011 Jul;301(1):E1-E10. doi: 10.1152/ajpendo.00667.2010. Epub 2011 Apr 12. PMID 21487075
- [Background] Zhang WY, Huang GY, Liu J. [Influences of acupuncture on infertility of rats with polycystic ovarian syndrome]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2009 Nov;29(11):997-1000. Chinese. PMID 20329610
- [Background] Stener-Victorin E, Waldenstrom U, Andersson SA, Wikland M. Reduction of blood flow impedance in the uterine arteries of infertile women with electro-acupuncture. Hum Reprod. 1996 Jun;11(6):1314-7. doi: 10.1093/oxfordjournals.humrep.a019378. PMID 8671446
- [Background] Manneras L, Jonsdottir IH, Holmang A, Lonn M, Stener-Victorin E. Low-frequency electro-acupuncture and physical exercise improve metabolic disturbances and modulate gene expression in adipose tissue in rats with dihydrotestosterone-induced polycystic ovary syndrome. Endocrinology. 2008 Jul;149(7):3559-68. doi: 10.1210/en.2008-0053. Epub 2008 Apr 3. PMID 18388196
- [Background] Zhao X, Ni R, Li L, Mo Y, Huang J, Huang M, Azziz R, Yang D. Defining hirsutism in Chinese women: a cross-sectional study. Fertil Steril. 2011 Sep;96(3):792-6. doi: 10.1016/j.fertnstert.2011.06.040. Epub 2011 Jul 18. PMID 21762890
- [Background] Ni RM, Mo Y, Chen X, Zhong J, Liu W, Yang D. Low prevalence of the metabolic syndrome but high occurrence of various metabolic disorders in Chinese women with polycystic ovary syndrome. Eur J Endocrinol. 2009 Sep;161(3):411-8. doi: 10.1530/EJE-09-0298. Epub 2009 Jun 19. PMID 19542239
- [Background] Chen X, Yang D, Li L, Feng S, Wang L. Abnormal glucose tolerance in Chinese women with polycystic ovary syndrome. Hum Reprod. 2006 Aug;21(8):2027-32. doi: 10.1093/humrep/del142. Epub 2006 May 9. PMID 16684838
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Cronin L, Guyatt G, Griffith L, Wong E, Azziz R, Futterweit W, Cook D, Dunaif A. Development of a health-related quality-of-life questionnaire (PCOSQ) for women with polycystic ovary syndrome (PCOS). J Clin Endocrinol Metab. 1998 Jun;83(6):1976-87. doi: 10.1210/jcem.83.6.4990. PMID 9626128
- [Background] Leung KF, Liu FB, Zhao L, Fang JQ, Chan K, Lin LZ. Development and validation of the Chinese Quality of Life Instrument. Health Qual Life Outcomes. 2005 Apr 16;3:26. doi: 10.1186/1477-7525-3-26. PMID 15833138
- [Background] Jiang M, Lu C, Zhang C, Yang J, Tan Y, Lu A, Chan K. Syndrome differentiation in modern research of traditional Chinese medicine. J Ethnopharmacol. 2012 Apr 10;140(3):634-42. doi: 10.1016/j.jep.2012.01.033. Epub 2012 Feb 1. PMID 22322251
- [Background] MacPherson H, Altman DG, Hammerschlag R, Youping L, Taixiang W, White A, Moher D; STRICTA Revision Group. Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA): extending the CONSORT statement. PLoS Med. 2010 Jun 8;7(6):e1000261. doi: 10.1371/journal.pmed.1000261. PMID 20543992
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Derived] Li J, Ng EH, Stener-Victorin E, Hu Z, Wu W, Lai M, Wu T, Ma H. Comparison of acupuncture pretreatment followed by letrozole versus letrozole alone on live birth in anovulatory infertile women with polycystic ovary syndrome: a study protocol for a randomised controlled trial. BMJ Open. 2016 Oct 7;6(10):e010955. doi: 10.1136/bmjopen-2015-010955. PMID 27855085